CLINICAL TRIAL: NCT02676583
Title: Effectiveness of Tonsil Fossa Closure in Pain Relief After Tonsillectomy in Children: Randomized Clinical Trial, Double-blind, Controlled Study
Brief Title: Effectiveness of Tonsil Fossa Closure in Pain Relief After Tonsillectomy in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Marco Aurelio Fornazieri (Other)
Collaborators: Universidade Estadual de Londrina (Other)
Responsible Party: Sponsor-Investigator, Marco Aurelio Fornazieri, Responsible MD, Clinica Olfact
Organization: Clinica Olfact (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: OLFACT-TONSIL-01
Record Dates: First submitted 2015-10-17; First posted 2016-02-08 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Tonsillitis
Keywords: pain; tonsillectomy; tonsillar fossa; suture; tonsil fossa closure
MeSH Terms: conditions — Tonsillitis; Pain | interventions — Tonsillectomy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Billateral tonsil fossa closure (Active Comparator): tonsillectomy
  Interventions: Procedure: Tonsillectomy
- No closure of tonsil fossa (Active Comparator): tonsillectomy
  Interventions: Procedure: Tonsillectomy
- Unilateral tonsil fossa closure (Active Comparator): tonsillectomy
  Interventions: Procedure: Tonsillectomy

INTERVENTIONS:
Procedure: Tonsillectomy — Closure or not closure of tonsil fossa

SUMMARY:
Objective: Postoperative pain is the main complaint in children undergoing tonsillectomy. An inexpensive method and with few evidence in the literature on effectiveness in reducing pain is the closure of the tonsillar fossa by suture with absorbable sutures. The investigators will compare the pain after tonsillectomy between closure or not the tonsil fossa.

Study design: Prospective, randomized, double blind, and controlled. Method: Two hundred otolaryngologic outpatients with indication of bilateral tonsillectomy for repeated tonsillitis, tonsillar hypertrophy or sleep apnea between 5 and 12 years old will be enrolled from November 2015 to July 2016. The procedure will be performed by a single surgeon and similar postoperative medications will be prescribed. There will be two techniques: closure or not of the tonsillar fossa with catgut points. A questionnaire containing a Faces Pain Scale - filled 1 and 7 days after surgery- and other data - difficulty of detachment of the palatine tonsils, hemostasis technique, surgical complications, healing characteristics, day of total improvement of the pain, day of beginning of normal food intake, presence of postoperative bleeding, complications and observations raised by the patient - will be applied.

ELIGIBILITY:
Inclusion Criteria:

* no cognitive-intellectual changes;
* capacity to respond the questionnaire;
* able to help in the study

Exclusion Criteria:

* conducting invasive procedure for less than two months;
* history of any infection during last month;
* continuous use of any medication;
* postoperative fever;
* non-standard medication prescribed for the postoperative time

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 131 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2017-07 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Pain | on post-operative procedure (1 day after surgery)
  Pain will be assessed using a questionnaire containing a Faces Pain Scale
Pain | on post-operative procedure (7 days after surgery)
  Pain will be assessed using a questionnaire containing a Faces Pain Scale. It will be evaluated the presence of the Pain and the change between the two time points as well.

SECONDARY OUTCOMES:
Resumption of normal diet | at 7 days after surgery
  wich day normal diet was recovered
Healing characteristics | at 7 days after surgery
  characteristics of edema, granuloma and uvula edema

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Olfact, Londrina, Paraná, Brazil